CLINICAL TRIAL: NCT03875274
Title: Postoperative Analgesic Effect of Morphine Added to Ropivacaine for Fascia Iliaca Compartment Block Following Femoral Fracture Surgeries
Brief Title: Morphine Added to Ropivacaine for FICB for Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Pankaj Baral, Junior Resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRC/0832/016
Record Dates: First submitted 2019-02-01; First posted 2019-03-14 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Morphine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine group (Placebo Comparator): Ropivacaine 0.375% 20 ml + Normal saline 2 ml via FICB
  Interventions: Drug: Ropivacaine, Saline
- Ropivacaine and morphine group (Experimental): Ropivacaine 0.375% 20 ml + Morphine 2 ml via FICB
  Interventions: Drug: Ropivacaine, Morphine

INTERVENTIONS:
Drug: Ropivacaine, Morphine — Morphine added to ropivacaine for fascia iliaca compartment block
  Arms: Ropivacaine and morphine group
Drug: Ropivacaine, Saline — Normal saline added to ropivacaine for fascia iliaca compartment block
  Arms: Ropivacaine group

SUMMARY:
prospective, randomized double blinded study to investigate the effects of morphine as an adjuvant to ropivacaine on FICB

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective femur surgery under spinal anaesthesia

  * Age group (18-65 years)
  * ASA physical status I and II

Exclusion Criteria:

* • Not willing to participate in the study

  * Other painful co-morbidities (neuropathies)
  * Allergy or any contraindication to study medication
  * Psychiatric disorder
  * Coagulopathy
  * Infection at the site of the block
  * Use of other modes of anaesthesia or analgesia besides spinal anaesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BPKIHS, Dharān, Sunsari, Nepal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine Group | Ropivacaine and Morphine Group
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Group | Ropivacaine and Morphine Group | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15) | 43 (12) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 20 | 25 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Nepal | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia
Description: The period in minutes when the patient is free of pain
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ropivacaine Group | Ropivacaine and Morphine Group
Number analyzed (Participants) | 35 | 35
minutes | 541 (167) | 634 (164)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Ropivacaine Group | Ropivacaine and Morphine Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03875274/Prot_SAP_ICF_000.pdf